CLINICAL TRIAL: NCT03280901
Title: HaemoDialysis Interventions to REduce Multi-Organ Dysfunction and Effect on Quality of Life (HD-REMODEL) Assessed by MRI Scanning
Brief Title: HaemoDialysis Interventions to REduce Multi-Organ Dysfunction and Effect on Quality of Life Assessed by MRI Scanning
Acronym: HD-REMODEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD-Remodel-UK-01; IRAS 207142 (Other Grant/Funding Number: Health Research Authority UK)
Record Dates: First submitted 2017-08-28; First posted 2017-09-13 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Renal Failure; Cardiovascular Diseases; Congenital Disorders
Keywords: renal replacement therapy; haemodialysis; haemodiafiltration
MeSH Terms: conditions — Renal Insufficiency; Cardiovascular Diseases; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: monocentric, block randomized, open, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard HD (Experimental): HD with constant temperature of 37°C, MRI scans of the heart, kidneys and brain during HD sessions
  Interventions: Other: HD, Magnetic Resonance Imaging (MRI) scans
- Thermocontrolled HD (Experimental): HD applying the Blood Temperature Monitor (BTM), MRI scans of the heart, kidneys and brain during HD sessions
  Interventions: Other: HD, Magnetic Resonance Imaging (MRI) scans

INTERVENTIONS:
Other: HD, Magnetic Resonance Imaging (MRI) scans — HD, Magnetic Resonance Imaging (MRI) scans using a specifically designed unit able to perform MRI scanning during HD sessions

SUMMARY:
The purpose of this study is to characterise in detail cardiac, cerebral and renal structure, function and perfusion in patients on haemodialysis (HD) using magnetic imaging techniques. The effects of a standard prescription haemodialysis (dialysate temperature 37 C) will be compared to a thermocontrolled (or isothermic) haemodialysis prescription to ascertain if thermocontrolled HD provides a protective effect on organ perfusion and circulatory stress when compared to conventional haemodialysis. The BTM (blood temperature monitor, Fresenius) offers a way to overcome this to regulate thermal balance during dialysis and achieve a neutral thermal balance (isothermic) over the dialysis session. Other dialysis parameters will be standardised between treatment arms using blood volume monitoring (BVM) and clinical assessments.

DETAILED DESCRIPTION:
The purpose of this study is to characterise in detail cardiac, cerebral and renal structure, function and perfusion in patients on haemodialysis (HD) using magnetic imaging techniques. The Primary objectives are to investigate the difference in cardiac perfusion, structure and function between standard HD and thermocontrolled HD using magnetic imaging techniques, to observe the the changes in renal perfusion and oxygenation within one dialysis session and the changes to cerebral perfusion within one dialysis session.

The secondary objectives are to investigate the difference in cerebral perfusion, structure, oedema and function between standard HD and thermocontrolled HD, the difference in renal perfusion and oxygenation between standard HD and thermocontrolled HD and the differences in visual acuity and cognitive assessment across a dialysis session and over a dialysis treatment course.

ELIGIBILITY:
Exclusion Criteria:

* Change in dry weight (clinically defined) in 4 weeks prior to recruitment
* Dialysate composition other than: sodium≥137mmol/L, potassium≥2.0mmol/L, calcium≥1.5mmol/L, magnesium≥0.5mmol/L, glucose 1.0g/L
* Instability on dialysis in 4 weeks prior to recruitment leading to either:

  * Emergency medical attention
  * Infusion of additional fluid
  * Loss in consciousness
  * Arrhythmia
  * Chest pain
  * Or any other medical condition that precludes the scan session in opinion of the investigator
* Dialysed via a synthetic line, central venous catheter or graft
* Qa < 500ml/min
* NYHA Stage IV heart failure (New York Heart Association)
* Active infection or malignancy
* Contraindication to MRI scanning including claustrophobia, pacemaker, metallic implants etc
* Pregnancy (pregnancy test will be conducted with female patients aged ≤ 55 years) or planning pregnancy or lactation period
* Medical conditions or overall physical frailty precludes scan session in opinion of investigator
* Unable or unwilling to provide informed consent
* Any condition which could interfere with the patient's ability to comply with the study
* Participation in an interventional clinical study during the preceding 30 days

Inclusion Criteria:

* Age 18-80, male and female
* Informed consent signed and dated by study patient and investigator/authorised physician
* Average (4 weeks prior to recruitment) Ultrafiltration volumes ≥ 0.5 litres/ dialysis session
* Receiving dialysis via an arteriovenous fistula
* Must be able to follow simple instruction in English (on safety grounds for MRI scans) and be able to understand the nature and requirements of the study
* Stable dialysis prescription
* CKD5 (Chronic kidney disease) patients having renal replacement therapy with haemodialysis/ haemodiafiltration (>90 days)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output during standard HD and thermocontrolled HD | after 2 and 4 weeks after randomisation
  Change in cardiac output during standard HD and thermocontrolled HD using Phase Contrast Magnetic Resonance Imaging (PC-MRI)
Change in renal perfusion during standard HD and thermocontrolled HD | after 2 and 4 weeks after randomisation
  Change in renal perfusion using Arterial Spin Labelling (ASL) and renal artery flow using PC-MRI
Change in cerebral perfusion during standard HD and thermocontrolled HD | after 2 and 4 weeks after randomisation
  Change in cerebral perfusion during standard HD and thermocontrolled HD using ASL

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, Professor, Study Chair — University of Nottingham, Division of Medical Sciences and Graduate Entry Medicine; Nicolas Selby, Dr, Principal Investigator — University of Nottingham, Division of Medical Sciences and Graduate Entry Medicine
Locations (1):
- University of Nottingham, Division of Medical Sciences and Graduate Entry Medicine, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No